CLINICAL TRIAL: NCT00001742
Title: The Role of Cyclooxygenase Activity in the Endothelial Function of Hypertensive and Hypercholesterolemic Patients
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980064; 98-H-0064
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-01

CONDITIONS: Healthy; Hypercholesterolemia; Hypertension
Keywords: Acetylcholine; Aspirin; Nitric Oxide; Sodium Nitroprusside; Hypercholesterolemia; Hypertension
MeSH Terms: conditions — Hypercholesterolemia; Hypertension

SUMMARY:
A layer of cells called the endothelium line the walls of blood vessels. These cells produce substances that control the tone of blood vessels and thus control blood flow through the vessel. This regulating activity of the endothelium is dysfunctional in several diseases of the heart and blood vessels, including high blood pressure and high levels of cholesterol.

Previous research has pointed toward a decrease in the action of nitric oxide (NO) as the cause of this abnormality. Nitric oxide is a substance produced by the cells of the endothelium that plays a role in the relaxation of blood vessels.

In this project researchers plan to study blood flow through the blood vessels in patients forearms after receiving four different drugs: sodium nitroprusside, acetylcholine, L-NMMA, and aspirin. These four drugs act on the blood vessels of the forearm through different mechanisms. Acetylcholine and sodium nitroprusside are drugs that open the blood vessels of the forearm and increase blood flow through the vessel. L-NMMA is a drug that blocks production of nitric oxide (NO). Aspirin's role in controlling blood flow is unknown.

Patients participating in this research study will not directly benefit from it. However, the study will contribute to researchers understanding of diseases of the blood vessels and heart.

DETAILED DESCRIPTION:
The endothelium modulates vascular tone by the release of constricting and relaxing substances that act on the underlying smooth muscle. This regulatory activity of the endothelium is dysfunctional in a number of cardiovascular conditions, including essential hypertension and hypercholesterolemia. Previous studies from our group have implicated a decreased action of endothelium-derived nitric oxide (NO) as the mechanism responsible for this abnormality. Whether this reduced bioactivity of NO is related to vasoactive prostanoids remains uncertain.

We propose to test the hypothesis that an increased production of vasoactive prostanoids by the cyclooxygenase (COX) system is responsible for the reduced bioactivity of NO in essential hypertension and hypercholesterolemia. We will investigate the effect of COX inhibition by aspirin (ASA) on resting vascular tone, and on both endothelium-dependent and independent vasodilation in normal subjects, hypertensive patients, and hypercholesterolemic patients.

For this purpose, we propose to analyze the regional vascular responses to acetylcholine (ACH) and to sodium nitroprusside (SNP) before and after the administration of ASA. We will also analyze the basal forearm blood flow (FBF) responses to increasing doses of ASA infusion. We will employ infusion of drugs into the brachial artery and we will measure the responses of the forearm vasculature by means of strain gauge plethysmography.

ELIGIBILITY:
Patients (men and nonpregnant women) with systemic hypertension and patients with hypercholesterolema will be included for this study.

Patient with aspirin allergies and those with a platelet count less than 50,000 will be excluded.

Volunteers cannot be in any kind of medication while participating in this study.

No history of diabetes, peripheral vascular disease, coagulopathy, or vasculitis.

Must be capable of rendering informed consent for all procedures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Start 1998-02; Study Completion 2001-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Moncada S, Vane JR. Pharmacology and endogenous roles of prostaglandin endoperoxides, thromboxane A2, and prostacyclin. Pharmacol Rev. 1978 Sep;30(3):293-331. No abstract available. PMID 116251
- [Background] Furchgott RF, Zawadzki JV. The obligatory role of endothelial cells in the relaxation of arterial smooth muscle by acetylcholine. Nature. 1980 Nov 27;288(5789):373-6. doi: 10.1038/288373a0. PMID 6253831
- [Background] Taddei S, Virdis A, Ghiadoni L, Magagna A, Salvetti A. Cyclooxygenase inhibition restores nitric oxide activity in essential hypertension. Hypertension. 1997 Jan;29(1 Pt 2):274-9. doi: 10.1161/01.hyp.29.1.274. PMID 9039114